CLINICAL TRIAL: NCT02742714
Title: Evaluation of PillCam SBC Capsule Endoscopy System Performance in Established and Suspected IBD Patients to Assess System Functionality by Visualizing and Assessing the Small Bowel and Colon
Brief Title: PillCam SBC System Functionality in Established and Suspected IBD Patients
Acronym: PIANO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: COVGIRD0546
Record Dates: First submitted 2016-03-02; First posted 2016-04-19 (Estimated); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Chronic Inflammatory Small Bowel Disease; Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PillCam SBC (Experimental): The PillCam SBC system to be tested in this study, is a new system composed of capsule, Data recorder and a new software Pillcam Desktop Software (version 9.0). The main features of the SBC capsule are panoramic field of view and adaptive frame rate customized for complete coverage of both small bowel and colonic mucosa.
  Interventions: Device: PillCam SBC system

INTERVENTIONS:
Device: PillCam SBC system — The PillCam SBC system to be tested in this study, is a new system composed of capsule, Data recorder and a new software Pillcam Desktop Software (version 9.0). The main features of the SBC capsule are panoramic field of view and adaptive frame rate customized for complete coverage of both small bowel and colonic mucosa.
  Other Names: PillCam Endoscopy system

SUMMARY:
This clinical study is designed to evaluate the PillCam SBC system performance in 50 established or suspected inflammatory bowel disease (IBD) patients by visualizing and assessing their small and large bowel.

DETAILED DESCRIPTION:
The PillCam SBC system to be tested in this study, is a new system composed of capsule, Data recorder and a new software Pillcam Desktop Software (version 9.0). The main features of the SBC capsule are panoramic field of view and adaptive frame rate customized for complete coverage of both small bowel and colonic mucosa.

Fifty established and suspected IBD patients (at least half of them with established crohn disease (CD)) with active or quiescent disease activity, aged 18 years and up, with no symptomatic stricture or known obstruction that would prevent capsule passage will be enrolled in up to 6 medical sites in Israel and Europe.

Patients will undergo bowel prep, followed by a PillCam SBC capsule examination. Patency capsule may precede PillCam SBC ingestion according to physician discretion.

The PillCam Software videos will be evaluated by local site reader following a Subjective Assessment Form fulfillment.

ELIGIBILITY:
Inclusion criteria:

* Patients ages 18-75 years, inclusive
* Patient has known crohn disease and/ or ulcerative colitis Or
* Patient suspected to have inflammatory bowel disease and suffers from either:
* Diarrhea for more than 6 weeks and/or
* Abdominal pain for more than 6 weeks and/or
* Extra-luminal manifestations of IBD including: erythema nodosum, pyoderma gangrenosum, arthritis, peri-anal disease, uveitis, aphthous stomatitis and
* Suffers from at least one of the symptoms / lab abnormalities listed below:

  * Positive inflammatory marker (ESR, C reactive protein (CRP), thrombocytosis, fecal lactoferrin, fecal calprotectin) within 3 months prior to enrollment
  * Unexplained anemia (less than normal limits) within 3 months prior to enrollment
  * Hypoalbuminemia (<3.5 g/dl) within 3 months of enrollment
  * Positive IBD serology within 3 months of enrollment
  * Recurrent Fevers
  * Unexplained weight loss
  * Gastro-intestinal bleeding including melena and/or hematochezia and/or fecal occult blood test (FOBT) positive.
  * Chronic perianal disease (fistula, fissure, peri-rectal abscess)
  * Abnormal imaging of Gastrointestinal (GI) tract (e.g. Magnetic resonance enterography (MRE)) suggestive of inflammatory bowel disease
* For known CD patients, proven patency by the patency capsule or another approach deemed clinically acceptable by the investigator, e.g. CT enterography, MRE performed within the 90 days prior to enrollment
* Patients agree to sign consent form

Exclusion criteria

* Antibiotic Associated Colitis
* Stool positive for Ova &Parasite and for Clostridium difficile toxin within 3 months of enrollment
* Other known infectious cause of symptoms
* Known or suspected intestinal obstruction
* Non-steroidal anti-inflammatory drugs (twice weekly or more) during the 4 weeks preceding enrollment.
* Suspected or known GI stricture, followed by patency capsule study or other imaging study that could not prove patency of the GI tract
* Patient is expected to undergo MRI examination within 7 days after ingestion of the capsule
* Patient with known gastrointestinal motility disorders
* Subjects with known or suspected delayed gastric emptying
* Patient suffers from any condition, such as swallowing problems, which precludes compliance with study and/or device instructions
* Patient has any allergy or other known contraindication or intolerance to the medications used in the study
* Patient has any condition, which precludes compliance with study and/or device instructions
* Women who are either pregnant or nursing at the time of screening, or are of child-bearing potential and do not practice medically acceptable methods of contraception
* Concurrent participation in another clinical trial using any investigational drug or device
* Patient suffers from a life threatening condition
* Patients with history or clinical evidence of renal disease and/or previous clinically significant laboratory abnormalities of renal function parameters

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-07; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Successful SBC procedure in terms of video creation and report generation per training instructions | 4 weeks
  Success procedures are being measured. Only if both video and report will be created it will be defined as success.

CONTACTS AND LOCATIONS:
Overall Officials: Abraham Eliakim, Prof., Principal Investigator — Sheba Medical Center
Locations (5):
- Israel (3):
  - Shaare Zedek Medical Center, Jerusalem
  - Sheba Medical Center, Ramat Gan
  - The Tel-Aviv Sourasky Medical Center, Tel Aviv
- Fondazione Policlinico Universitario Agostino Gemelli, Rome, Italy
- Hospital de Navarra, Pamplona, Spain

IPD SHARING:
Plan to Share IPD: No